CLINICAL TRIAL: NCT01068886
Title: External Pancreatic Duct Stent After Pancreaticoduodenectomy: a Prospective Randomized Multicenter Trial
Brief Title: External Pancreatic Duct Stent After Pancreaticoduodenectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Yvonnick MORICE, Centre Hospitalier Universitaire
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC 04-04
Record Dates: First submitted 2005-09-14; First posted 2010-02-15 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Pancreatic Fistula
Keywords: Pancreaticoduodenectomy
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no stent (No Intervention): no stent through pancreatic anastomosis
- stent (Experimental): stent through pancreatic anastomosis
  Interventions: Procedure: External pancreatic stent

INTERVENTIONS:
Procedure: External pancreatic stent — stent through pancreatic anastomosis
  Other Names: pancreatic stent
  Arms: stent

SUMMARY:
Pancreatoduodenectomy (PD) is performed in many high volume centers with a very low mortality. Reduced mortality rate is largely the result of careful patient selection, improved intraoperative management and a better postoperative care. Unfortunately, there is not a similar reduction in morbidity rates which remains about 40%. Persistent morbidity is predominantly due to pancreatic fistula (PF). Abdominal abscess and hemorrhage are common sequelae of PF which have been associated with a high mortality rate. While many different risk factors have been reported, a soft pancreatic texture and a nondilated pancreatic duct have been most consistently linked to high rates of PF. A number of methods for reducing the incidence of PF have been proposed and analysed. Many of these involve technical features of the anastomosis, including site of reconstruction, anastomotic technique, use of biologic glue, and prophylactic use of somatostatin analogue. The placement of a stent through the pancreatic anastomosis is an attractive strategy to reduce the PF rate. This multicenter prospective randomized trial was designed to compare the outcome after PD with external drainage stent versus no stent in patients with high risk of PF (with soft pancreas and a diameter of wirsung <3mm).

Analysis:The primary objective of the study was to compare the incidence PF in patients with or without external pancreatic stent. With an anticipated PF rate of 30%, based on literature experience, it was calculated that a reduction to 10% of PF rate would require the inclusion of 75 patients in each group (statistical significance P < 0.05 and power 80 per cent with a two-tailed test of proportions). We'll enroll 158 patients to take into account the possibility of 5% being lost to follow-up.

DETAILED DESCRIPTION:
Analysis: The primary objective of the study was to compare the incidence PF in patients with or without external pancreatic stent. With an anticipated PF rate of 30%, based on literature experience, it was calculated that a reduction to 10% of PF rate would require the inclusion of 75 patients in each group (statistical significance P < 0.05 and power 80 per cent with a two-tailed test of proportions). We'll enroll 158 patients to take into account the possibility of 5% being lost to follow-up.

PF was defined, according to the International Study Group of Pancreatic Fistula, as amylase rich fluid (amylase concentration more than three times serum concentration) collected from the drainage placed intraoperatively from day 3 or by needle aspiration of an intraabdominal collection. PF were graded according to the clinical impact on the patient's hospital course (grades A,B,C).

ELIGIBILITY:
Inclusion criteria:

* All patients scheduled for elective PD,
* Confirmation of the soft pancreas or nondilated pancreatic duct during PD.

Exclusion criteria:

* Age less than 18 year,
* Emergency surgery,
* Previous pancreatic surgery,
* Previous susmesocolic radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-01; Primary Completion 2009-04 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
pancreatic fistula | on postoperative day 30

SECONDARY OUTCOMES:
overall morbidity | postoperative day 30

CONTACTS AND LOCATIONS:
Overall Officials: arnaud - jean-pierre, professor, Principal Investigator — University Hospital
Locations (1):
- University Hospital, Angers, France

REFERENCES:
- [Derived] Pessaux P, Sauvanet A, Mariette C, Paye F, Muscari F, Cunha AS, Sastre B, Arnaud JP; Federation de Recherche en Chirurgie (French). External pancreatic duct stent decreases pancreatic fistula rate after pancreaticoduodenectomy: prospective multicenter randomized trial. Ann Surg. 2011 May;253(5):879-85. doi: 10.1097/SLA.0b013e31821219af. PMID 21368658